CLINICAL TRIAL: NCT07026708
Title: Target Investigation of Residual Inflammation After Non-ST/ ST Elevation Acute Coronary Syndrome - TIRANA (ACS) Prospective REGISTRY
Brief Title: TIRANA-ACS: A Prospective Registry Study for the Targeted Investigation of Residual Inflammation After Non-ST/ ST Elevation Acute Coronary Syndrome
Acronym: TIRANA (ACS)
Status: Recruiting | Type: Observational
Sponsor: University Hospital Centre Mother Teresa (Other)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: 3232
Record Dates: First submitted 2025-06-10; First posted 2025-06-18 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: ACS (Acute Coronary Syndrome); Myocardial Infarction (MI); Myocardial Inflammation; Inflammation Biomarkers; NSTEMI - Non-ST Segment Elevation MI; STEMI
Keywords: Residual inflammation; Myocardial infarction; Percutaneous Coronary Intervention; Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Myocarditis; Non-ST Elevated Myocardial Infarction; ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute Coronary Syndrome Patients: Data Collection:
  General patient information, diagnosis, comorbidities, CRP levels, neutrophil and lymphocyte counts, thrombocyte count, HDL cholesterol, LDL cholesterol, and complications (electrical and mechanical) will be collected from the medical records in the cardiology department of our main tertiary hospital "Mother Teresa Hospital".
  Angiographic data and treatment information will be gathered from standard coronary angiography reports used at our cardiac catheterization laboratories.
  The follow-up form used for telephone interviews with patients is based on standardized instruments, including the WHO Rose Angina Questionnaire, Seattle Angina Questionnaire, EQ-5D-5L, MacNew Heart Disease Health-Related Quality of Life Questionnaire, McGill Pain Questionnaire, and the MRC Dyspnoea Scale.
  Patient status will be evaluated at 24 hours, 48 hours, and 6 months after the onset of symptoms. The symptom onset time will be obtained from medical records documented upon patient referral.

SUMMARY:
This prospective observational study aims to evaluate the prognostic significance of the neutrophil-to-lymphocyte ratio (NLR) as a predictor of mortality in patients following an episode of Acute Coronary Syndrome (ACS). Despite advancements in interventional cardiology and medical therapy, mortality remains significant in post-ACS patients, and early risk stratification is essential for optimizing outcomes.

Recent studies have suggested that systemic inflammatory markers, such as NLR, are associated with adverse cardiovascular events. It is an easily obtainable and cost-effective laboratory parameter derived from a routine complete blood count. However, its value as an independent predictor of mortality post-ACS has not yet been fully established in our population.

The study will include patients aged, admitted with a confirmed diagnosis of ACS (STEMI or Non-STEMI) and treated with percutaneous coronary intervention (PCI). NLR values will be measured from the first blood draw upon hospital admission, 24 and 48 hours post PCI. Patients will be followed up for up to 6 months after discharge through telephone interviews .

First, primary outcomes of the study will be the association between NLR values and mortality (all cause mortality and cardiovascular mortality), MACE (MACE was defined as the composite of all-cause mortality, cardiac death, unplanned revascularization, non-fatal myocardial infarction that was attributable and not related to stent failure or unplanned revascularization not related to stent failure) within 6 months post-ACS.

Secondary outcomes will include:

1. Differences in mean NLR between STEMI and NSTEMI patients.
2. Association between elevated NLR and the presence of multivessel coronary artery disease on angiography.
3. Correlation of NLR with other biomarkers, including the platelet-to-lymphocyte ratio (PLR), C-reactive protein (CRP), high-density lipoprotein (HDL) cholesterol, and maximum troponin levels (as an indicator of myocardial infarction size)

This study aims to contribute to the identification of easily accessible and cost-efficient biomarkers that can aid clinicians in early risk stratification of ACS survivors. A strong correlation between high NLR values and increased post-discharge mortality would suggest that inflammation plays a key role in patient prognosis and could potentially influence post-ACS management strategies.

ELIGIBILITY:
Inclusion Criteria:

- All patients (undergoing PCI, aged 18-85 years) presenting to the cardiology department or/and the cardiology intensive care unit with a diagnosis of ACS

Exclusion Criteria:

* Patients presenting to the cardiology department or/and the cardiology intensive care unit with diagnoses other than ACS and/or UA. Patients who died before undergoing PCI and those who did not provide a contact number.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General patient information, diagnosis, comorbidities, CRP levels, neutrophil and lymphocyte counts, thrombocyte count, HDL cholesterol, LDL cholesterol, and complications (electrical and mechanical) will be collected from the medical records in the cardiology department of our main tertiary hospital "Mother Teresa Hospital".
  Angiographic data and treatment information will be gathered from standard coronary angiography reports used at our cardiac catheterization laboratories.
  The follow-up form used for telephone interviews with patients is based on standardized instruments, including the WHO Rose Angina Questionnaire, Seattle Angina Questionnaire, EQ-5D-5L, MacNew Heart Disease Health-Related Quality of Life Questionnaire, McGill Pain Questionnaire, and the MRC Dyspnoea Scale.
  Patient status will be evaluated at 24 hours, 48 hours, and 6 months after the onset of symptoms. The symptom onset time will be obtained from medical records documented upon patient referral.
Sampling Method: Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Neutrophil-to-Lymphocyte Ratio (NLR) | 6 months post-ACS with a potential prolonged period of roughly 12 months
  Association Between Neutrophil-to-Lymphocyte Ratio (NLR) and Mortality (all cause mortality and cardiovascular mortality), MACE (MACE was defined as the composite of all-cause mortality, cardiac death, unplanned revascularization, non-fatal myocardial infarction that was attributable and not related to stent failure or unplanned revascularization not related to stent failure) in Post-Acute Coronary Syndrome (ACS) Patients .
  This outcome assesses the predictive value of NLR levels for mortality within 6 months following an ACS event.
Mortality (all cause mortality and cardiovascular mortality) | 6 months post-ACS with a potential prolonged period of roughly 12 months
  Mortality (all cause mortality and cardiovascular mortality) in Post-Acute Coronary Syndrome (ACS) Patients .
MACE (Major Acute Coronary Events) | 6 months post-ACS with a potential prolonged period of roughly 12 months
  MACE was defined as the composite of all-cause mortality, cardiac death, unplanned revascularization, non-fatal myocardial infarction that was attributable and not related to stent failure or unplanned revascularization not related to stent failure in Post-Acute Coronary Syndrome (ACS) Patients .

SECONDARY OUTCOMES:
Difference in Mean NLR Between STEMI and NSTEMI Patients | At hospital admission
  This outcome evaluates the variation in mean NLR values among patients diagnosed with ST-Elevation Myocardial Infarction (STEMI) versus Non-ST-Elevation Myocardial Infarction (NSTEMI).
  Time Frame: At hospital admission
Association Between High NLR and Presence of Multivessel Coronary Artery Disease | During initial coronary angiography
  This outcome explores whether elevated NLR values are associated with the presence of multivessel disease identified during coronary angiography.
Correlation Between NLR and Other Inflammatory Markers (PLR, CRP, HDL-Cholesterol) | Within 48 hours of hospital admission
  This outcome assesses the relationship between the NLR and other laboratory markers of inflammation and cardiovascular risk, including platelet-to-lymphocyte ratio (PLR), C-reactive protein (CRP), and HDL-cholesterol levels.
Correlation Between NLR and Peak Troponin Levels | During hospitalization (within first 5 days of admission)
  This outcome evaluates the correlation between baseline NLR and peak troponin levels as a surrogate marker for myocardial infarction size.

CONTACTS AND LOCATIONS:
Overall Officials: Andi Rroku, MD, Principal Investigator — Deutsches Herzzentrum der Charité (DHZC) - Campus Benjamin Franklin; Alban Dibra, Prof. Dr, Phd, Study Director — University of Medicine, Tirana; Martiola Kola, MD, Principal Investigator — University of Medicine, Tirana
Locations (1):
- Faculty of Medicine Tirana, Tirana, Albania

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT07026708/Prot_SAP_000.pdf
  • Informed Consent Form (2025-06-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT07026708/ICF_001.pdf